CLINICAL TRIAL: NCT04135001
Title: Mental Flexibility Study
Brief Title: Mental Flexibility
Acronym: MFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: WRAIR #2686
Record Dates: First submitted 2019-09-25; First posted 2019-10-22 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Anger; Hostility

STUDY DESIGN:
Intervention Model Description: Assignment to each condition (active vs. placebo) will be done by block assignment (by company) using the two versions of the HBMT program start code by study staff running participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBM Training (Experimental)
  Interventions: Behavioral: HBM Training
- Placebo Training (Placebo Comparator)
  Interventions: Other: Placebo Training

INTERVENTIONS:
Behavioral: HBM Training — A computer-based training to reduce hostile bias and interpersonal conflict as a mechanism to improve trust and cohesion within an operational military unit across the deployment cycle. The computer training is based on the Go/No-Go task (Fillmore et al., 2006) and Lexical Decision Task (Lepore & Brown, 2002). The training reduces HAB by affecting two cognitive mechanisms: prime seeking non-hostile concepts when presented with ambiguous cues and conditioning inhibition in response to hostile cues. Thus, the training induces a non-hostile attribution bias while simultaneously training the inhibition of hostile attribution bias and aggressive behavior in response to ambiguous cues.
  Arms: HBM Training
Other: Placebo Training — Volunteers in the placebo condition will be told to complete the fragments with the first word that comes to mind. This placebo still exposes volunteers to the training stimuli and computer task, but does not train inhibition or selectively prime non-hostility, which are the hypothesized mechanisms of the training.
  Arms: Placebo Training

SUMMARY:
The main purpose of this research is evaluate if HBMT reduces HAB in Soldiers, reduces intra-team conflict, improves trust, and improves unit cohesion. A secondary purpose of this research is to test Soldier acceptability and perception of the training. Volunteers will be randomized to a training or placebo version of a computer task designed to reduce HAB and interpersonal conflict. Soldiers will then complete surveys at multiple time intervals before, during, and following deployment. If successful, this research would demonstrate the ability of a computer based training to improve unit cohesion and Soldier attitudes during pre-deployment training and deployment itself.

DETAILED DESCRIPTION:
The study will consist of a double blind randomized controlled trial of HBMT (versus placebo) with subsequent pre-, during, and post-deployment surveys to assess the effectiveness of HBMT to influence relevant unit- and Soldier-level outcomes. Soldiers will be Command directed to participate. As such, all data will be used for briefing to unit leadership, however, participants will be asked to consent whether they allow their data to be used for research purposes. Subordinate units within the BN will be randomly assigned to complete either an active training or placebo version of the task. The individual briefing the Soldiers during training sessions will not know which version of the training the Soldiers are completing on the computer. Up to 40 Soldiers will complete HBMT at a time on individual study computers. Brief surveys will follow each training. There will also be a survey shortly before deployment, during deployment and shortly after deployment. See Appendix Q for tentative study timeline. For details on procedure see Section 9.8. Surveys completed during same day as HBMT training sessions will be completed on experimenter provided laptops, whereas surveys completed independent of an HBMT training session will be completed in pencil and paper format. See section 219.8 for details. The current protocol provides details for the first time point (initial HBMT training session). Additional amendments will be used to provide details and obtain approval for subsequent time points as these are coordinated with the unit. However, general information for follow-on time points is provided in this version of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Soldiers assigned to the 1-128 IN BN / Wisconsin Army National Guard.

Exclusion Criteria:

* Soldiers not assigned to the 1-128 IN BN / Wisconsin Army National Guard.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2023-08-06 (Estimated); Study Completion 2024-08-06 (Estimated)

PRIMARY OUTCOMES:
attitudes about mission | throughout study to completion, up to 1 year
  Attitudes toward Mission. Nine items based on past WRAIR research that assess Soldiers attitudes about their mission.
Workplace interpersonal conflict scale | throughout study to completion, up to 1 year
  Workplace Interpersonal Conflict Scale. Adapted from Wright et al., 2017
unit cohesion measure | throughout study to completion, up to 1 year
  Three item measure used in past WRAIR research. Based on Podsakoff and MacKenzie (1994)

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: No